CLINICAL TRIAL: NCT04050150
Title: Task-oriented Training of Arm Function in Standing After Stroke: a Pilot Study
Brief Title: Arm Training in Standing After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Jill Stewart, PT, PhD, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080332
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Stroke
Keywords: Rehabilitation; Upper Extremity
MeSH Terms: conditions — Stroke | interventions — Standing Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm Training in Standing (Experimental): Task-oriented, functional arm training completed in standing or during walking. All participants receive the same arm training intervention.
  Interventions: Behavioral: Arm training in standing

INTERVENTIONS:
Behavioral: Arm training in standing — Arm training will be provided in one hour sessions, 3 time per week for 8 weeks. In each session, you will practice functional tasks with your weaker arm and hand in standing or during walking. Practice will be scaled to match your current level of function and progressed over time as able.

SUMMARY:
This study will examine the feasibility of providing task-oriented arm training in standing or during walking in individuals with movement deficits due to stroke. Participants will received 24 sessions of arm training in standing over an 8-week period that focus on arm and hand function.

DETAILED DESCRIPTION:
Residual motor deficits are common after stroke and often have a negative impact on the performance of functional activities and overall quality of life. A frequently reported contribution to these functional limitations is an inability to incorporate the weaker arm and hand into daily activities. While rehabilitation interventions can improve arm functional capacity, these improvements often do not translate into increased real-world arm use which is often reduced after stroke.

The performance of skilled arm and hand movements in standing requires precise coordination between upper extremity movement and balance control. Many everyday functional tasks that require the arm are performed in standing (e.g. opening a door or meal preparation at the kitchen counter), however, training of arm function in rehabilitation is often done in sitting. An important rehabilitation approach may be to create a training environment that resembles the way the arm is used in everyday life (i.e. standing). This study will examine the feasibility of providing task-oriented, functional arm training in standing and during walking in individuals with motor deficits due to stroke.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Had a stroke at least 6 months prior to enrollment
* Show evidence of continued arm and hand weakness
* Have some ability to move the arm and hand that is weaker from the stroke
* Be able to stand with minimal assistance or less without support of the weaker arm for at least 2 minutes
* Be able to follow two-step commands.

Exclusion Criteria:

* Acute medical issues that would interfere with participation
* Another neurologic diagnosis that may impact movement (e.g. Parkinson's Disease)
* Severe apraxia or hemispatial neglect
* Pain that interferes with arm movement or standing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Sessions Completed | 8 weeks
  Total number of treatment sessions completed
Fatigue | 8 weeks
  Mean change in self-reported fatigue from the start to the end of each intervention session
Treatment intensity | 8 weeks
  Total number of arm repetitions per session and the percent of arm repetitions completed in standing or walking
Action Research Arm Test | Change from Baseline to 8 weeks
  Clinical measure of arm and hand function
Arm Use Measured with Accelerometers | Change from Baseline to 8 weeks
  Arm use measured during a typical day using accelerometers worn on the wrist

SECONDARY OUTCOMES:
Upper Extremity Fugl-Meyer | Change from Baseline to 8 weeks
  Clinical Measure of arm and hand impairment
Box & Blocks Test | Change from Baseline to 8 weeks
  Clinical measure of hand function
Nine-Hole Peg Test | Change from Baseline to 8 weeks
  Clinical measure of hand dexterity
Stroke Impact Scale Hand Domain Subscale | Change from Baseline to 8 weeks
  Patient-reported measure of hand related quality-of-life. Score ranges from 0 to 100 with higher being better.
Timed Up and Go | Change from Baseline to 8 weeks
  Clinical measure of mobility and balance
Activities Specific Balance Confidence Scale | Change from Baseline to 8 weeks
  Patient-reported measure of balance confidence. Score ranges from 0 to 100 with higher being better

OTHER OUTCOMES:
Berg Balance Scale | Change from Baseline to 8 weeks
  Clinical measure of balance. 14-item performance measure with a maximum score of 56; higher score is better.
Functional Gait Assessment | Change from Baseline to 8 weeks
  Clinical measure of balance
Stroke Impact Scale Mobility Subscale | Change from Baseline to 8 weeks
  Patient-reported measure of mobility related quality-of-life. Score ranges from 0 to 100 with higher being better
Action Research Arm Test | Change from Baseline to 12 weeks
  Clinical measure of arm and hand function
Arm Use Measured with Accelerometers | Change from Baseline to 12 weeks
  Arm use measured during a typical day using accelerometers worn on the wrist

CONTACTS AND LOCATIONS:
Overall Officials: Jll Stewart, PT, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available per reasonable request to the principal investigator 1 year after study completion.
Time Frame: 1 year after study completion